CLINICAL TRIAL: NCT03669146
Title: The Enhancement Via Accommodation (EVA) Study
Brief Title: Enhancement of Emmetropization in Highly Hyperopic Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donald O Mutti, OD, PhD (Other)
Responsible Party: Sponsor-Investigator, Donald O Mutti, OD, PhD, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEW-33235
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Hyperopia
Keywords: Emmetropization; Refractive Error; Glasses; Accommodation
MeSH Terms: conditions — Hyperopia; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: A provider other than the investigator(s) will be masked to the primary outcome of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Hyperopic subjects receiving glasses (Experimental): Randomized +5.00 to +7.00 diopter hyperopic subjects that will receive partial refractive correction and will be instructed to do accommodation exercises on a daily basis.
  Interventions: Device: Glasses
- Hyperopic subjects uncorrected (No Intervention): Randomized +5.00 to +7.00 diopter hyperopic subjects that will serve as the control to the experimental arm who will receive no correction but be observed for the duration of the study.
- Highly hyperopic subjects corrected (Active Comparator): If a subject is found to be greater than +7.00 diopters hyperopic during the screening phase of the study, they will receive glasses correction and be followed during the study period.
  Interventions: Device: Glasses

INTERVENTIONS:
Device: Glasses — Partial refractive correction in a pair of glasses.
  Arms: Highly hyperopic subjects corrected; Hyperopic subjects receiving glasses

SUMMARY:
Infants do not usually wear glasses because they usually do not need them to see clearly. Most infants are born with a moderate amount of farsightedness. Most infants then undergo a natural process called 'emmetropization' that reduces the amount of farsightedness. However, up to 10% of infants don't emmetropize and end up with very farsighted prescriptions. Farsighted infants must use extra focusing effort to see clearly, which may make their eyes cross and perhaps cause a "lazy eye". If infants avoid this effort and their vision stays blurred into childhood, they may develop two lazy eyes. Farsightedness in school-aged children makes reading and learning more difficult. New studies in animals and in humans show that infant eyes will emmetropize best if they have just a normal, moderate amount of farsightedness. The infant eye must be in this normal target zone in order to emmetropize. If a baby were given glasses with the full prescription to correct all of his farsightedness, the eyes would also be out of the target zone and would not receive any signal to grow. The best strategy might be to give a partial spectacle correction for the farsightedness, just enough to put them in the zone that is most effective for emmetropization.

The purpose of this project is to determine if emmetropization can be enhanced in very farsighted babies. We will give them glasses with a partial correction and accommodative (eye focusing) training. The partial correction is an amount that is less than their full degree of farsightedness but enough to put them in the zone of effective emmetropization. As changes in farsightedness occur, the power of the glasses will be reduced to keep the farsightedness within the target zone. If an infant reaches a normal amount of farsightedness, the glasses will be discontinued. The comparison group will be farsighted babies who receive the current standard of care, namely no correction. The main outcome of the study will be whether there is a significant difference in the decrease of farsightedness between the two groups when the infants are 18 months of age.

If emmetropization can be enhanced in very farsighted babies, the risk of developing crossed or lazy eye will be reduced. The lifelong need for spectacles, contact lenses, or refractive surgery for high amounts of farsightedness would also be reduced. Positive results might also make infant eye examinations more common and place a new therapeutic option in clinicians' hands.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 8 and 15 weeks at baseline examination
* Either gender
* Any ethnicity
* Birthweight greater than 2500g
* Normal pregnancy and delivery (including Cesarean section delivery but excluding serious complications or conditions such as eclampsia or rubella)
* Hyperopia greater than or equal to +5.00 Diopters (D) in the spherical component of refractive error in one or both eyes measured with cycloplegic retinoscopy using 1% cyclopentolate
* Infants with a refractive error of greater than or equal to +5.00D but less than or equal to +7.00D in the spherical component of refractive error will be randomized to treatment (partial correction with accommodative training) or observation only.
* Infants with greater than +7.00D in the spherical component of refractive error will receive treatment

Exclusion Criteria:

* Astigmatism greater than 2.00D in either eye
* Anisometropia greater than 1.50D (spherical equivalent)
* History of strabismus surgery
* History of difficulty with pupillary dilation
* History of cardiac, liver, asthma, or other respiratory disease
* History of ocular disease, retinal detachment, severe macular dragging, intraocular surgery, optic nerve hypoplasia, malformations of the eye, cortical visual impairment or active inflammation
* History of hydrocephalus, Down syndrome, cerebral palsy, developmental delay, seizure disorders

Ages: 8 Weeks to 15 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald O Mutti, OD, PhD, Principal Investigator — Ohio State University; Ann M Morrison, OD, PhD, Study Chair — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morrison AM, Robich ML, Jordan LA, Sinnott LT, Mutti DO. Emmetropization in highly hyperopic infants: A randomized clinical trial of partial refractive correction. Optom Vis Sci. 2025 May 1;102(5):310-319. doi: 10.1097/OPX.0000000000002254. Epub 2025 Apr 10. PMID 40261678
- [Derived] Morrison AM, Mutti DO. Evaluation of a Pilot Protocol for Detecting Infant Hyperopia. Optom Vis Sci. 2023 May 1;100(5):304-311. doi: 10.1097/OPX.0000000000002011. Epub 2023 Mar 23. PMID 36951871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperopic Subjects Receiving Glasses | Hyperopic Subjects Uncorrected | Highly Hyperopic Subjects Corrected
Started | 15 | 15 | 5
Completed | 13 | 14 | 5
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperopic Subjects Receiving Glasses | Hyperopic Subjects Uncorrected | Highly Hyperopic Subjects Corrected | Total
Number analyzed (Participants) | 15 | 15 | 5 | 35
Age, Continuous [Mean (Standard Deviation); unit: Days] | 81.9 (10.2) | 79.0 (9.0) | 78.6 (8.7) | 80.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 4 | 20
  Male | 6 | 8 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 5 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 14 | 15 | 4 | 33
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Central Cycloplegic Refractive Error With Retinoscopy
Description: The subject's central refractive error will be measured (in Diopters) with cycloplegic retinoscopy to determine if partial refractive correction and accommodative training can enhance emmetropization in highly hyperopic infants. Successful enhancement is defined as being an average of 1.75 Diopters less hyperopic than control subjects at 18 months.
Time Frame: 18 months
Population: Subject numbers here do not match initial projected subject numbers due to participant drop outs (2 in hyperopic subjects receiving glasses; 1 in hyperopic subjects uncorrected)
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Pairs of eyes
Arm/Group | Hyperopic Subjects Receiving Glasses | Hyperopic Subjects Uncorrected | Highly Hyperopic Subjects Corrected
Number analyzed (Participants) | 13 | 14 | 5
Number analyzed (Pairs of eyes) | 13 | 14 | 5
Diopters | 1.6 (0.6) | 1.2 (0.7) | 2.8 (1.2)

2. Secondary Outcome: Peripheral Cycloplegic Refractive Error With SureSight Autorefractor
Description: The subject's central and peripheral refractive error will be measured (in Diopters) with the SureSight autorefractor to determine if partial refractive correction and accommodative training can enhance emmetropization through modulation of ocular shape in highly hyperopic infants.
Time Frame: 18 months
Population: Number analyzed is slightly less due to drop outs of participants (2 in treatment/hyperopic subjects with glasses; 1 observation/uncorrected no glasses)
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Pairs of eyes
Arm/Group | Hyperopic Subjects Receiving Glasses | Hyperopic Subjects Uncorrected | Highly Hyperopic Subjects Corrected
Number analyzed (Participants) | 13 | 14 | 5
Number analyzed (Pairs of eyes) | 13 | 14 | 5
Diopters
  Central Spherical Equivalent Refractive Error | 2.15 (0.61) | 1.99 (1.18) | 4.11 (1.11)
  Relative Nasal Spherical Equivalent Refractive Error | -0.28 (0.89) | -0.19 (0.6) | -0.52 (0.25)
  Relative Temporal Spherical Equivalent Refractive Error | -1.25 (1.17) | -0.81 (0.77) | -2.21 (0.61)

3. Secondary Outcome: Accommodative Response With PowerRefractor
Description: The subject's accommodative ability will be measured objectively with a PowerRefractor autorefractor to determine determine if partial refractive correction and accommodative training can enhance emmetropization through modulation of accommodation in highly hyperopic infants.
Time Frame: 18 months
Population: Final number analyzed slightly less due to participant drop out (2 in treatment/hyperopic subjects receiving glasses and 1 observation/hyperopic subjects uncorrected)
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Pairs of eyes
Arm/Group | Hyperopic Subjects Receiving Glasses | Hyperopic Subjects Uncorrected | Highly Hyperopic Subjects Corrected
Number analyzed (Participants) | 13 | 14 | 5
Number analyzed (Pairs of eyes) | 13 | 14 | 5
Diopters | 2.21 (0.00) | 2.09 (0.22) | 1.97 (0.23)

ADVERSE EVENTS:
Time Frame: 15 months
Description: All-Cause Mortality: No participants in the study died Serious Adverse Events: No participants developed any serious adverse events Other (Not Including Serious) Adverse Events: No adverse events reported from participants
Arm/Group | Hyperopic Subjects Receiving Glasses | Hyperopic Subjects Uncorrected | Highly Hyperopic Subjects Corrected
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/5

LIMITATIONS AND CAVEATS:
Small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT03669146/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT03669146/ICF_001.pdf